CLINICAL TRIAL: NCT07071246
Title: Rituximab for the Treatment of New-onset AChR-Myasthenia Gravis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202206-13
Record Dates: First submitted 2022-07-12; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Treatment
Keywords: myasthenia gravis; rituximab; efficacy; safety
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RTX intravenously for the treatment of myasthenia gravis (Other): RTX administrating 100mg per week consecutively for 3 weeks
  Interventions: Drug: Rituximab Injection

INTERVENTIONS:
Drug: Rituximab Injection — low dose of rituximab intravenously
  Other Names: RTX

SUMMARY:
Myasthenia gravis (MG) is the most common acquired disorder of neuromuscular junction (NMJ), the most common antibody (in 85% MG patients) being the nicotinic acetylcholine receptor (AChR). Traditional medical treatments of new-onset MG include anticholinesterase inhibitors, immunomodulating therapies such as intravenous immunoglobulin (IVIG) and plasma exchange (PLEX) and immunosuppressive agents such as corticosteroids, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate and cyclophosphamide. Since a status of complete stable remission (CSR, defined as remission of MG without pharmacological treatment≥1 year) is difficult to achieve, the international consensus guidance for management of MG proposed "minimal manifestation (MM) or better status" with no greater than mild adverse events as a practical goal of MG treatment. Given the balance between efficacy and safety, a more aggressive strategy and approach for immune therapies are critical in early stage of new-onset MG. In clinical practice, biological agent monoclonal antibody rituximab (RTX), specifically targeting B-lymphocyte differentiation membrane antigen CD20, has been increasing in recent years for some immune-mediated neurological diseases such as multiple sclerosis (MS) and neuromyelitis optica spectrum disorders (NMOSD), and gradually represented potential advantages in immunosuppressive therapy-refractory and new-onset AChR-MG. However, up to now, the individualized regimen, optimal dosage and clinical benefit of RTX monotherapy for early stage of new-onset AChR-MG still need to be elucidated. This study was performed to assess the long-term clinical efficacy and safety of individualized low-dose 100 mg RTX monotherapy approach in new-onset AChR-MG patients.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is the most common acquired disorder of neuromuscular junction (NMJ), in which pathogenic autoantibodies bind to components of the postsynaptic membrane in NMJ, the most common antibody (in 85% MG patients) being the nicotinic acetylcholine receptor (AChR), followed by muscle-specific kinase (MuSK) or lipoprotein related peptide 4 (LRP4), thereby making impairment of neuromuscular transmission, causing fatigable weakness and even representing a potentially life-threatening condition. Traditional medical treatments of new-onset MG include anticholinesterase inhibitors such as pyridostigmine for temporarily symptomatic relief, immunomodulating therapies such as intravenous immunoglobulin (IVIG) and plasma exchange (PLEX) for a rapid but short-term clinical response, and immunosuppressive agents such as corticosteroids, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate and cyclophosphamide for long-term treatment. Moreover, accompanied with prolonged duration, approximately 20% of the generalized MG population develop to refractory progressive course even with long-time and sufficient traditional immunosuppressive agents. For all newly diagnosed MG patients, chest computed tomography (CT) scan must be performed to assess for thymoma, and thymectomy should be done immediately in those thymoma patients with IVIG or PLEX treatment 1 to 2 weeks prior to thymectomy for optimizing condition, then followed by additional medical therapy for a sustained disease control. Since a status of complete stable remission (CSR, defined as remission of MG without pharmacological treatment≥1 year) is difficult to achieve, the international consensus guidance for management of MG proposed "minimal manifestation (MM) or better status" with no greater than mild adverse events as a practical goal of MG treatment. Given the balance between efficacy and safety, a more aggressive strategy and approach for immune therapies are critical in early stage of new-onset MG. AChR-MG is an archetype for B cell-mediated autoimmune disorder, clearly implicating a principal role for B cells in the disease pathogenesis. Therefore, B lymphocytes have always been the focus of investigative interests, especially with the successful introduction of biological therapeutics that target these cells. In clinical practice, biological agent monoclonal antibody rituximab (RTX), specifically targeting B-lymphocyte differentiation membrane antigen CD20, has been increasing in recent years for some immune-mediated neurological diseases such as multiple sclerosis (MS) and neuromyelitis optica spectrum disorders (NMOSD), and gradually represented potential advantages in immunosuppressive therapy-refractory and new-onset AChR-MG. However, up to now, the individualized regimen, optimal dosage and clinical benefit of RTX monotherapy for early stage of new-onset AChR-MG still need to be elucidated. This study was performed to assess the long-term clinical efficacy and safety of individualized low-dose 100 mg RTX monotherapy approach in new-onset AChR-MG patients, using MG Foundation of America (MGFA)-Postintervention Status (PIS) "Minimal Manifestation (MM) or better status" as the primary outcome, changes in Quantitative Myasthenia Gravis (QMG), Manual Muscle Testing (MMT), MG-Related Activities of Daily Living (MG-ADL), and 15-item Quality-of-Life (MGQOL-15) scores as the secondary outcomes, as well as cholinesterase inhibitors reduction, peripheral CD19+B-cell percentage, AChR antibody titers and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the informed consent form, and the subjects were willing to complete the research protocol as planned;
2. The age is over 18 years old, and the gender is not limited (women of childbearing age have a negative pregnancy test);
3. Meet the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Myasthenia Gravis (2020 Edition);
4. The subjects of the study are all Chinese Han people;
5. Good physical condition;
6. Complete demographic and clinical data during the baseline survey and follow-up;
7. Serum AChR antibody positive;
8. New-onset AChR-MG, with symptoms no more than 12 months;
9. American Myasthenia Gravis Foundation (MGFA) clinical classification grades I to IV (grade I only indicates ocular muscle weakness, grade II mild systemic disease, grade III moderate systemic disease, grade IV severe systemic disease , Grade V requires intubation crisis);
10. The patient has never received immunosuppressive therapy or RTX therapy. If receiving cortisol hormone therapy, the oral dose should be less than 3 months, and the daily dose should not exceed 40 mg.

Exclusion Criteria:

1. Myasthenic crisis at screening (MGFA grade V);
2. Accompanied with serious physical diseases, such as severe heart failure;
3. Liver and kidney insufficiency or elevated transaminases (AST/ALT elevation exceeds 2.5 times the upper limit of normal)
4. Suffering from clinical depression symptoms and serious mental illness;
5. Combined with other neurological diseases, with a history of organic brain diseases and traumatic brain injury;
6. Use of immunosuppressive agents, including rituximab, azathioprine, mycophenolate mofetil, cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus or methotrexate, etc.;
7. Potential acute or chronic viral or bacterial infection, such as HIV, latent hepatitis B, tuberculosis, etc.;
8. Vaccination history within 4 weeks before enrollment;
9. During pregnancy or breastfeeding;
10. Those who cannot sign the informed consent;
11. Patients with poor compliance;
12. Any other situation in which the investigator believes that the patient should not participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
70% enrolled patients reached the minimum state (MM) or better state of MGFA - post intervention state (PIs) at 1 year after administration of study drug | 12 months
  No functional impairment and some muscle weakness may be detected by a specialist neurologist
80% enrolled patients reached the clinical complete remission (CSR) of MGFA - post intervention status (PIs) at 2 years after administration of study drug | 24 months
  No signs and symptoms of muscle weakness for at least 1 year, no medical treatment for MG during this period, no evidence of muscle weakness after examination by a professional neurologist, mild eyelid closure weakness is allowed
Safety: The incidence of treatment-related adverse reactions and withdrawal because of serious adverse reaction | through study completion
  Any adverse reaction, like fever, rash, dizziness and so on.

SECONDARY OUTCOMES:
The proportion of patients with ocular myasthenia gravis (OMG) progressed to generalized myasthenia gravis (GMG). | After 2 years of follow-up
  OMG progressed to the GMG at 2 years after treatment of study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016 Dec 29;375(26):2570-2581. doi: 10.1056/NEJMra1602678. No abstract available. PMID 28029925
- [Background] Morren J, Li Y. Maintenance immunosuppression in myasthenia gravis, an update. J Neurol Sci. 2020 Mar 15;410:116648. doi: 10.1016/j.jns.2019.116648. Epub 2019 Dec 26. PMID 31901719
- [Background] Rath J, Brunner I, Tomschik M, Zulehner G, Hilger E, Krenn M, Paul A, Cetin H, Zimprich F. Frequency and clinical features of treatment-refractory myasthenia gravis. J Neurol. 2020 Apr;267(4):1004-1011. doi: 10.1007/s00415-019-09667-5. Epub 2019 Dec 11. PMID 31828474
- [Background] Mantegazza R, Antozzi C. From Traditional to Targeted Immunotherapy in Myasthenia Gravis: Prospects for Research. Front Neurol. 2020 Sep 2;11:981. doi: 10.3389/fneur.2020.00981. eCollection 2020. PMID 32982957
- [Background] Sanders DB, Wolfe GI, Benatar M, Evoli A, Gilhus NE, Illa I, Kuntz N, Massey JM, Melms A, Murai H, Nicolle M, Palace J, Richman DP, Verschuuren J, Narayanaswami P. International consensus guidance for management of myasthenia gravis: Executive summary. Neurology. 2016 Jul 26;87(4):419-25. doi: 10.1212/WNL.0000000000002790. Epub 2016 Jun 29. PMID 27358333
- [Background] Jaretzki A 3rd, Barohn RJ, Ernstoff RM, Kaminski HJ, Keesey JC, Penn AS, Sanders DB. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology. 2000 Jul 12;55(1):16-23. doi: 10.1212/wnl.55.1.16. No abstract available. PMID 10891897
- [Background] Brauner S, Eriksson-Dufva A, Hietala MA, Frisell T, Press R, Piehl F. Comparison Between Rituximab Treatment for New-Onset Generalized Myasthenia Gravis and Refractory Generalized Myasthenia Gravis. JAMA Neurol. 2020 Aug 1;77(8):974-981. doi: 10.1001/jamaneurol.2020.0851. PMID 32364568
- [Background] Di Stefano V, Lupica A, Rispoli MG, Di Muzio A, Brighina F, Rodolico C. Rituximab in AChR subtype of myasthenia gravis: systematic review. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):392-395. doi: 10.1136/jnnp-2019-322606. Epub 2020 Feb 25. PMID 32098874
- [Background] Punga AR, Maddison P, Heckmann JM, Guptill JT, Evoli A. Epidemiology, diagnostics, and biomarkers of autoimmune neuromuscular junction disorders. Lancet Neurol. 2022 Feb;21(2):176-188. doi: 10.1016/S1474-4422(21)00297-0. PMID 35065040
- [Background] Huijbers MG, Marx A, Plomp JJ, Le Panse R, Phillips WD. Advances in the understanding of disease mechanisms of autoimmune neuromuscular junction disorders. Lancet Neurol. 2022 Feb;21(2):163-175. doi: 10.1016/S1474-4422(21)00357-4. PMID 35065039
- [Background] Uzawa A, Kuwabara S, Suzuki S, Imai T, Murai H, Ozawa Y, Yasuda M, Nagane Y, Utsugisawa K. Roles of cytokines and T cells in the pathogenesis of myasthenia gravis. Clin Exp Immunol. 2021 Mar;203(3):366-374. doi: 10.1111/cei.13546. Epub 2020 Dec 3. PMID 33184844
- [Background] Villegas JA, Bayer AC, Ider K, Bismuth J, Truffault F, Roussin R, Santelmo N, Le Panse R, Berrih-Aknin S, Dragin N. Il-23/Th17 cell pathway: A promising target to alleviate thymic inflammation maintenance in myasthenia gravis. J Autoimmun. 2019 Mar;98:59-73. doi: 10.1016/j.jaut.2018.11.005. Epub 2018 Dec 18. PMID 30578016
- [Background] Li Y, Guptill JT, Russo MA, Howard JF Jr, Massey JM, Juel VC, Hobson-Webb LD, Emmett D, Chopra M, Raja S, Liu W, Yi JS. Imbalance in T follicular helper cells producing IL-17 promotes pro-inflammatory responses in MuSK antibody positive myasthenia gravis. J Neuroimmunol. 2020 Aug 15;345:577279. doi: 10.1016/j.jneuroim.2020.577279. Epub 2020 May 27. PMID 32497931
- [Background] Yilmaz V, Maillard S, Truffault F, Bolgert F, Behin A, Regnard JF, Berrih-Aknin S, Le Panse R. Regulatory B cells in myasthenia gravis are differentially affected by therapies. Ann Clin Transl Neurol. 2018 Sep 22;5(11):1408-1414. doi: 10.1002/acn3.645. eCollection 2018 Nov. PMID 30480034
- [Background] Bergantini L, d'Alessandro M, Cameli P, Vietri L, Vagaggini C, Perrone A, Sestini P, Frediani B, Bargagli E. Effects of rituximab therapy on B cell differentiation and depletion. Clin Rheumatol. 2020 May;39(5):1415-1421. doi: 10.1007/s10067-020-04996-7. Epub 2020 Feb 22. PMID 32088800
- [Background] Forsthuber TG, Cimbora DM, Ratchford JN, Katz E, Stuve O. B cell-based therapies in CNS autoimmunity: differentiating CD19 and CD20 as therapeutic targets. Ther Adv Neurol Disord. 2018 Mar 21;11:1756286418761697. doi: 10.1177/1756286418761697. eCollection 2018. PMID 29593838
- [Background] Dos Santos A, Noury JB, Genestet S, Nadaj-Pakleza A, Cassereau J, Baron C, Videt D, Michel L, Pereon Y, Wiertlewski S, Magot A. Efficacy and safety of rituximab in myasthenia gravis: a French multicentre real-life study. Eur J Neurol. 2020 Nov;27(11):2277-2285. doi: 10.1111/ene.14391. Epub 2020 Jul 4. PMID 32526053
- [Background] Singh N, Goyal V. Rituximab as induction therapy in refractory myasthenia gravis: 18 month follow-up study. J Neurol. 2019 Jul;266(7):1596-1600. doi: 10.1007/s00415-019-09296-y. Epub 2019 Mar 27. PMID 30919039
- [Background] Choi K, Hong YH, Ahn SH, Baek SH, Kim JS, Shin JY, Sung JJ. Repeated low-dose rituximab treatment based on the assessment of circulating B cells in patients with refractory myasthenia gravis. Ther Adv Neurol Disord. 2019 Sep 18;12:1756286419871187. doi: 10.1177/1756286419871187. eCollection 2019. PMID 31555344
- [Background] Li H, Huang Z, Jia D, Xue H, Pan J, Zhang M, Shi K, Shi FD, Zhang C. Low-dose rituximab treatment for new-onset generalized myasthenia gravis. J Neuroimmunol. 2021 May 15;354:577528. doi: 10.1016/j.jneuroim.2021.577528. Epub 2021 Feb 24. PMID 33662696
- [Background] Zhang C, Bu B, Yang H, Wang L, Liu W, Duan RS, Zhang M, Zeng P, Du C, Yang L, Shi FD. Immunotherapy choice and maintenance for generalized myasthenia gravis in China. CNS Neurosci Ther. 2020 Dec;26(12):1241-1254. doi: 10.1111/cns.13468. Epub 2020 Oct 26. PMID 33103369
- [Background] Li T, Zhang GQ, Li Y, Dong SA, Wang N, Yi M, Qi Y, Zhai H, Yang L, Shi FD, Yang CS. Efficacy and safety of different dosages of rituximab for refractory generalized AChR myasthenia gravis: A meta-analysis. J Clin Neurosci. 2021 Mar;85:6-12. doi: 10.1016/j.jocn.2020.11.043. Epub 2021 Jan 2. PMID 33581791
- [Background] Lu J, Zhong H, Jing S, Wang L, Xi J, Lu J, Zhou L, Zhao C. Low-dose rituximab every 6 months for the treatment of acetylcholine receptor-positive refractory generalized myasthenia gravis. Muscle Nerve. 2020 Mar;61(3):311-315. doi: 10.1002/mus.26790. Epub 2020 Jan 6. PMID 31875994
- [Background] Anderson D, Phan C, Johnston WS, Siddiqi ZA. Rituximab in refractory myasthenia gravis: a prospective, open-label study with long-term follow-up. Ann Clin Transl Neurol. 2016 May 25;3(7):552-5. doi: 10.1002/acn3.314. eCollection 2016 Jul. PMID 27386504
- [Background] Robeson KR, Kumar A, Keung B, DiCapua DB, Grodinsky E, Patwa HS, Stathopoulos PA, Goldstein JM, O'Connor KC, Nowak RJ. Durability of the Rituximab Response in Acetylcholine Receptor Autoantibody-Positive Myasthenia Gravis. JAMA Neurol. 2017 Jan 1;74(1):60-66. doi: 10.1001/jamaneurol.2016.4190. PMID 27893014
- [Background] Du Y, Li C, Hao YF, Zhao C, Yan Q, Yao D, Li L, Zhang W. Individualized regimen of low-dose rituximab monotherapy for new-onset AChR-positive generalized myasthenia gravis. J Neurol. 2022 Aug;269(8):4229-4240. doi: 10.1007/s00415-022-11048-4. Epub 2022 Mar 3. PMID 35243555